CLINICAL TRIAL: NCT03519932
Title: A Bilateral Dispensing Comparison of Biofinity Toric and Ultra for Astigmatism
Brief Title: Comparison of Comfilcon A Toric Contact Lenses and Samfilcon A Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-91
Record Dates: First submitted 2018-05-01; First posted 2018-05-09 (Actual); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- comfilcon A toric lens (Experimental): Subjects who wear comfilcon A toric lens either as first or second pair during this cross-over study.
  Interventions: Device: comfilcon A toric lens; Device: samfilcon A toric lens
- samfilcon A toric lens (Active Comparator): Subjects who wear samfilcon A toric lens either as first or second pair during this cross-over study.
  Interventions: Device: comfilcon A toric lens; Device: samfilcon A toric lens

INTERVENTIONS:
Device: comfilcon A toric lens — Contact lens
  Other Names: Biofinity toric; test lens
Device: samfilcon A toric lens — Contact lens
  Other Names: Ultra for Astigmatism; control lens

SUMMARY:
The objective of this study is to evaluate the subjective acceptance of comfilcon A toric contact lens, compared to samfilcon A toric lens.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer;
* Has had a self-reported oculo-visual examination in the last two years.
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Is an adapted soft contact lens wearer, who currently wears contact lenses for a minimum 3 days/week and 8 hours/day AND who anticipates no difficulty wearing CLs for 6 days/week, 10 hours /day.
* Is willing to wear contact lens in both eyes for the duration of the study;
* Has a minimum astigmatism of - 0.75, determined by refraction;
* Can be fit with the two study contact lens types in the powers available;
* Has a distance visual acuity of 0.20 logMAR (approx 20/30) or better, determined by refraction;
* Can achieve a distance visual acuity of 0.20 logMAR (approx 20/30) or better in each eye with the study contact lenses.
* Has clear corneas and no active* ocular disease

Exclusion Criteria:

* Is participating in any concurrent clinical trial;
* Has any known active* ocular disease and/or infection;
* Has a systemic condition that in the opinion of the investigator may affect a study measure;
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study measure;
* Has known sensitivity to fluorescein dye or products to be used in the study;
* Appears to have any active* ocular pathology, ocular anomaly or severe insufficiency of lacrimal secretion (severe dry eye) that would affect the wearing of contact lenses;
* Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
* Is aphakic;
* Has undergone refractive error surgery.
* Has participated in the PIANO (i.e. EX-MKTG-83) Study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Principal Investigator — Director, Centre for Ocular Research & Education
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized to wear comfilcon A toric lenses for 1-month and samfilcon A toric lenses for 1-month in this cross-over dispensing study.
Groups:
- Comfilcon A Toric Then Samfilcon A Toric: Subjects were randomized to wear comfilcon A toric lenses for 1-month and then crossover to wear Samfilcon A toric lenses for 1-month.
  Contact Lens: comfilcon A toric Contact Lens: Samfilcon A toric
- Samfilcon A Toric Then Comfilcon A Toric: Subjects were randomized to wear sammfilcon A toric lenses for 1-month and then crossover to wear comfilcon A toric lenses for 1-month.
  Contact Lens: Samfilcon A toric Contact Lens: comfilcon A toric
Period: First Intervention
Arm/Group | Comfilcon A Toric Then Samfilcon A Toric | Samfilcon A Toric Then Comfilcon A Toric
Started | 24 | 25
Completed | 23 (One subject had non-significant adverse event and data not included in the analysis) | 22 (3 subjects had non-significant adverse events and data not included in analysis.)
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 3
Period: Second Intervention
Arm/Group | Comfilcon A Toric Then Samfilcon A Toric | Samfilcon A Toric Then Comfilcon A Toric
Started | 22 (Subjects who wore samfilcon A toric at 1st intervention wear comfilcon A toric at 2nd intervention) | 23 (Subjects who wore comfilcon A toric at 1st intervention wear Samfilcon A toric at 2nd intervention)
Completed | 22 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 49

OUTCOME MEASURES:

1. Primary Outcome: Comfort at Insertion
Description: Subjective ratings of comfort for each pair of lenses (scale: 0-10; 0=painful,10=can't feel lens)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A Toric Lens: Subjects were randomized to wear comfilcon A toric lens and samfilcon A toric lens during this cross-over study.
  comfilcon A toric lens: Contact lens
- Samfilcon A Toric Lens: Subjects were randomized to wear samfilcon A toric lens and comfilcon A toric lens during this cross-over study.
  samfilcon A toric lens: Contact lens
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 45 | 45
units on a scale | 9.0 (1.2) | 8.8 (1.2)

2. Primary Outcome: Comfort
Description: Subjective ratings of comfort for each pair of lenses (scale: 0-10; 0=painful,10=can't feel lens)
Time Frame: 2 weeks
Population: One subject's subjective rating was excluded for comfilcon A toric due to subject confusion at rating scale and potentially reversing its use.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 44 | 45
units on a scale
  Overall | 8.1 (1.4) | 7.4 (2.1)
  Removal | 7.2 (2.1) | 6.5 (2.4)

3. Primary Outcome: Comfort
Description: Subjective ratings of comfort for each pair of lenses (scale: 0-10; 0=painful,10=can't feel lens)
Time Frame: 1-month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 45 | 44
units on a scale
  Overall | 8.1 (1.6) | 7.4 (2.1)
  Removal | 7.1 (2.1) | 6.7 (2.5)

4. Primary Outcome: Lens Preference Based on Overall Comfort
Description: Lens preference with respect to comfort (Prefer pair-1 strongly, Prefer pair-1 slightly, Prefer pair-2 strongly, prefer pair-2 slightly, No preference)
Time Frame: 1 month
Population: Percentages may be rounded and therefore may not add up to equal to 100%
Measure: Number; unit: percentage of participants
Groups:
- Overall Preference: Subjects were randomized to wear comfilcon A toric lens and samfilcon A toric lens during this cross-over study for a month.
  comfilcon A toric lens: Contact lens
  samfilcon A toric lens: Contact lens
Arm/Group | Overall Preference
Number analyzed (Participants) | 45
percentage of participants
  Strongly prefer comfilcon A | 44
  Slightly Prefer comfilcon A | 27
  No Preference | 7
  Slightly prefer samfilcon A | 7
  Strongly prefer samfilcon A | 16

5. Primary Outcome: Lens Preference Based on Overall Dryness
Description: Lens preference with respect to dryness (Prefer pair-1 strongly, Prefer pair-1 slightly, Prefer pair-2 strongly, prefer pair-2 slightly, No preference)
Time Frame: 1 month
Measure: Number; unit: percentage of participants
Groups:
- Overall Participants: Subjects were randomized to wear comfilcon A toric lens and samfilcon A toric lens during this cross-over study for a month.
  comfilcon A toric lens: Contact lens
  samfilcon A toric lens: Contact lens
Arm/Group | Overall Participants
Number analyzed (Participants) | 45
percentage of participants
  Strongly prefer comfilcon A | 29
  Slightly prefer comfilcon A | 33
  No Preference | 16
  Slightly prefer samfilcon A | 4
  Strongly prefer samfilcon A | 18

6. Primary Outcome: Dryness
Description: Subjective ratings of dryness for each pair of lenses (scale: 0-10; 0=Extremely dry, 10=No dryness)
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 44 | 45
units on a scale
  Overall | 7.4 (2.0) | 6.9 (2.2)
  Removal | 6.5 (2.5) | 6.0 (2.3)

7. Primary Outcome: Dryness
Description: Subjective ratings of dryness for each pair of lenses (scale: 0-10; 0=Extremely dry, 10=No dryness)
Time Frame: 1-month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A Toric Lens: Subjects were randomized to wear comfilcon A toric lens and samfilcon A toric during this cross-over study.
  comfilcon A toric lens: Contact lens
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 45 | 45
units on a scale
  Overall | 7.5 (1.8) | 6.7 (2.5)
  Removal | 6.6 (2.3) | 6.2 (2.6)

8. Secondary Outcome: Ease of Insertion
Description: Subjective rating of ease of inserting the lens onto the eye (scale 0-10; 0=very difficult, 10=very easy)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 45 | 45
units on a scale | 9.3 (1.0) | 9.3 (0.9)

9. Secondary Outcome: Ease of Insertion
Description: Subjective rating of ease of inserting the lens onto the eye (scale 0-10; 0=very difficult, 10=very easy)
Time Frame: 2-weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 44 | 45
units on a scale | 8.9 (1.5) | 8.4 (1.9)

10. Secondary Outcome: Ease of Insertion
Description: Subjective rating of ease of inserting the lens onto the eye (scale 0-10; 0=very difficult, 10=very easy)
Time Frame: 1-month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 45 | 45
units on a scale | 9.0 (1.4) | 8.3 (1.8)

11. Secondary Outcome: Ease of Removal
Description: Subjective rating of ease of removing the lens from the eye (scale 0-10; 0=very difficult, 10=very easy)
Time Frame: 2-weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 44 | 45
units on a scale | 7.9 (2.5) | 8.4 (1.8)

12. Secondary Outcome: Ease of Removal
Description: Subjective rating of ease of removing the lens from the eye (scale 0-10; 0=very difficult, 10=very easy)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Toric Lens | Samfilcon A Toric Lens
Number analyzed (Participants) | 45 | 45
units on a scale | 8.0 (2.4) | 8.5 (1.7)

ADVERSE EVENTS:
Time Frame: One month during each crossover period.
Groups:
- Comfilcon A Toric: Subjects were randomized to wear comfilcon A toric lenses for 1-month and samfilcon A toric lenses for 1-month in this cross-over dispensing study.
  Contact Lens: comfilcon A toric
- Samfilcon A Toric: Subjects were randomized to wear samfilcon A toric lenses for 1-month and comfilcon A toric lenses for 1-month in this cross-over dispensing study.
  Contact Lens: samfilcon A toric
Arm/Group | Comfilcon A Toric | Samfilcon A Toric
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT03519932/Prot_SAP_000.pdf